CLINICAL TRIAL: NCT05534724
Title: Is Full Weight Bearing After the Modified Lapidus Operation Possible? A Randomized Controlled Trial to Compare Early and Partial Weight-bearing
Brief Title: A Study to Compare Early and Partial Weight-bearing After Hallux Valgus Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORL-ORT-033
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Hallux Valgus; Orthopedic Disorder
Keywords: Quality of life; Bone consolidation; Foot surgery; Lapidus surgery; Weil surgery; Hohmann surgery; Akin surgery
MeSH Terms: conditions — Hallux Valgus; Musculoskeletal Diseases | interventions — Partial Weight-Bearing

STUDY DESIGN:
Intervention Model Description: The surgical operation will be the modified Lapidus arthrodesis of hallux valgus with/without an Akin or a Weil/Hohmann surgery fusion.
  Post-operatively, patients will be randomized into one of the two groups:
  * Group A (control intervention): immediate post-operative partial weight-bearing (10 - 15kg) with a VACOPASO for 6 weeks, crutches and antithrombotic prophylaxis.
  * Group B (experimental intervention): immediate post-operative complete weight-bearing with a VACOPASO for 6 weeks and antithrombotic prophylaxis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial weight-bearing (10 - 15kg) (Other): Immediate post-operative partial weight-bearing (10 - 15kg) with a VACOPASO shoe for 6 weeks, crutches and antithrombotic prophylaxis
  Interventions: Other: Partial weight-bearing (10 - 15kg)
- Complete weight-bearing (Experimental): Immediate post-operative complete weight-bearing with a VACOPASO shoe for 6 weeks and antithrombotic prophylaxis
  Interventions: Other: Complete weight-bearing

INTERVENTIONS:
Other: Partial weight-bearing (10 - 15kg) — Immediate post-operative partial weight-bearing (10 - 15kg) with a VACOPASO shoe for 6 weeks
  Arms: Partial weight-bearing (10 - 15kg)
Other: Complete weight-bearing — Complete post-operative weight-bearing with a VACOPASO shoe for 6 weeks
  Arms: Complete weight-bearing

SUMMARY:
This is a two-arm randomized controlled trial with the aim to evaluate the effectiveness and safety of post-operative management after a modified Lapidus arthrodesis with/without an Akin or a Weil/Hohmann surgery fusion with immediate complete weight-bearing compared with partial weight-bearing (10 - 15kg) for 6 weeks as a novel approach for rehabilitation after a foot surgery.

DETAILED DESCRIPTION:
The surgical operation will be carried out according to the standard clinical practice, namely following the modified Lapidus general and specific rules concerning the surgical treatment of hallux valgus with/without an Akin or a Weil/Hohmann surgery fusion. Post-operatively, patients who meet the eligibility criteria will be randomized into one of the two groups (partial weight-bearing limited at 15kg vs full weight-bearing) Patient in both groups will be wearing a VACOPASO shoe for 6 weeks.

Standard X-ray assessment to determine healing, hardware fixation, fracture alignment, fracture reduction, implants mobilization will be performed at weeks 6, 12, 24.

Change in pain severity from the day of surgery to 6, 12 and 24 weeks postoperatively will be measured using the pain Visual Analogue Scale (VAS). Quality of life will be assessed through the American Orthopedic Foot and Ankle Score (AOFAS). Subjective functional recovery through the Olerud and Molander Ankle Score (OMAS).

ELIGIBILITY:
Inclusion Criteria:

* Patient who undergo modified Lapidus arthrodesis operation and associated with:
* Additional surgical gestures such as e.g. interventions on the proximal phalanx of the first finger (Akin) or interventions on the 2nd and / or 3rd ray (Weil / Hohmann) [23,24].
* Willingness and ability to participate in the trial
* Signed Informed Consent

Exclusion Criteria:

* Diabetes mellitus
* Rheumatoid arthritis
* Previous foot surgery
* Classic Lapidus surgery
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, general physical problem of the participant, etc.
* Inability or contraindications to undergo the investigated intervention
* Pregnant women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Subjective functional recovery measured by Olerud and Molander Ankle Score (OMAS) | at 6 weeks
  The Olerud and Molander Ankle Score (OMAS) is a functional rating scale from 0 to 100 and is based on nine different items: pain, stiffness, swelling, stair climbing, running, jumping, squatting, supports and activities of daily living. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Pain on a Visual Analogue Scale | At the day of surgery, at 6, 12 and 24 weeks postoperatively.
  Change in pain severity postoperatively measured using the pain Visual Analogue Scale (VAS).
  The pain VAS scale is a validated, self-assessment scale in which patients rate their pain by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (0) and "worst pain" (10).
Bone consolidation through anteroposterior and lateral foot x-rays | 6 weeks and 12 weeks. At 24 weeks in case of fracture non-union reported at the 12th week postoperatively
  Incidence of bone consolidation (bone callus formation) assessed in an objective measure by the radiologist
American Orthopedic Foot and Ankle Score questionnaire | at 6, 12 and 24 weeks
  The American Orthopedic Foot and Ankle Score (AOFAS) is used find the quality of life index for foot-and-ankle pathologies. It is made of nine questions and cover three categories: Pain (40 points), function (50 points) and alignment (10 points). These are all scored together for a total of 100 points. Higher scores mean a better outcome.
Subjective functional recovery measured by Olerud and Molander Ankle Score (OMAS) | at 12 and 24 weeks
  Subjective functional recovery through the Olerud and Molander Ankle Score (OMAS).
  The Olerud and Molander Ankle Score (OMAS) [7] is a functional rating scale from 0 to 100 and is based on nine different items: pain, stiffness, swelling, stair climbing, running, jumping, squatting, supports and activities of daily living. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Riegger, MD, Principal Investigator — EOC
Locations (1):
- EOC, Lugano, Switzerland

REFERENCES:
- [Background] Olerud C, Molander H. A scoring scale for symptom evaluation after ankle fracture. Arch Orthop Trauma Surg (1978). 1984;103(3):190-4. doi: 10.1007/BF00435553. PMID 6437370
- [Background] LAPIDUS PW. A quarter of a century of experience with the operative correction of the metatarsus varus primus in hallux valgus. Bull Hosp Joint Dis. 1956 Oct;17(2):404-21. No abstract available. PMID 13413410
- [Background] Butson AR. A modification of the Lapidus operation for hallux valgus. J Bone Joint Surg Br. 1980 Aug;62(3):350-2. doi: 10.1302/0301-620X.62B3.6997319.
- [Result] Kitaoka HB, Alexander IJ, Adelaar RS, Nunley JA, Myerson MS, Sanders M. Clinical rating systems for the ankle-hindfoot, midfoot, hallux, and lesser toes. Foot Ankle Int. 1994 Jul;15(7):349-53. doi: 10.1177/107110079401500701. PMID 7951968
- [Result] Drummond D, Motley T, Kosmopoulos V, Ernst J. Stability of Locking Plate and Compression Screws for Lapidus Arthrodesis: A Biomechanical Comparison of Plate Position. J Foot Ankle Surg. 2018 May-Jun;57(3):466-470. doi: 10.1053/j.jfas.2017.10.025. Epub 2018 Feb 19. PMID 29472168
- [Result] Ray RG, Ching RP, Christensen JC, Hansen ST Jr. Biomechanical analysis of the first metatarsocuneiform arthrodesis. J Foot Ankle Surg. 1998 Sep-Oct;37(5):376-85. doi: 10.1016/s1067-2516(98)80045-8. PMID 9798168
- [Result] Sangeorzan BJ, Hansen ST Jr. Modified Lapidus procedure for hallux valgus. Foot Ankle. 1989 Jun;9(6):262-6. doi: 10.1177/107110078900900602. PMID 2744666
- [Result] Myerson M, Allon S, McGarvey W. Metatarsocuneiform arthrodesis for management of hallux valgus and metatarsus primus varus. Foot Ankle. 1992 Mar-Apr;13(3):107-15. doi: 10.1177/107110079201300301. PMID 1601337
- [Result] Bednarz PA, Manoli A 2nd. Modified lapidus procedure for the treatment of hypermobile hallux valgus. Foot Ankle Int. 2000 Oct;21(10):816-21. doi: 10.1177/107110070002101004. PMID 11128011
- [Result] Saxena A, Nguyen A, Nelsen E. Lapidus bunionectomy: Early evaluation of crossed lag screws versus locking plate with plantar lag screw. J Foot Ankle Surg. 2009 Mar-Apr;48(2):170-9. doi: 10.1053/j.jfas.2008.12.009. PMID 19232969
- [Result] Blitz NM, Lee T, Williams K, Barkan H, DiDimenico LA. Early weight bearing after modified lapidus arthodesis: a multicenter review of 80 cases. J Foot Ankle Surg. 2010 Jul-Aug;49(4):357-62. doi: 10.1053/j.jfas.2010.04.014. PMID 20610203
- [Result] Kopp FJ, Patel MM, Levine DS, Deland JT. The modified Lapidus procedure for hallux valgus: a clinical and radiographic analysis. Foot Ankle Int. 2005 Nov;26(11):913-7. doi: 10.1177/107110070502601103. PMID 16309603
- [Result] Catanzariti AR, Mendicino RW, Lee MS, Gallina MR. The modified Lapidus arthrodesis: a retrospective analysis. J Foot Ankle Surg. 1999 Sep-Oct;38(5):322-32. doi: 10.1016/s1067-2516(99)80003-9. PMID 10553545
- [Result] Myerson MS, Badekas A. Hypermobility of the first ray. Foot Ankle Clin. 2000 Sep;5(3):469-84. PMID 11232392
- [Result] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Result] Arnold H. [The Akin procedure as closing wedge osteotomy for the correction of a hallux valgus interphalangeus deformity]. Oper Orthop Traumatol. 2008 Dec;20(6):477-83. doi: 10.1007/s00064-008-1503-8. German. PMID 19137394
- [Result] Podskubka A, Stedry V, Kafunek M. [Distal shortening osteotomy of the metatarsals using the Weil technique: surgical treatment of metatarsalgia and dislocation of the metatarsophalangeal joint]. Acta Chir Orthop Traumatol Cech. 2002;69(2):79-84. Czech. PMID 12073646
- [Result] Christensen PH, Hansen TB. Hallux valgus correction using a modified Hohmann technique. Foot Ankle Int. 1995 Apr;16(4):177-80. doi: 10.1177/107110079501600401. PMID 7787972
- [Result] Nix S, Smith M, Vicenzino B. Prevalence of hallux valgus in the general population: a systematic review and meta-analysis. J Foot Ankle Res. 2010 Sep 27;3:21. doi: 10.1186/1757-1146-3-21. PMID 20868524
- [Result] Deal JB Jr, Patzkowski JC, Groth AT, Ryan PM, Dowd TC, Osborn PM, Anderson CD, Ficke JR, Kirk KL. Early vs Delayed Weightbearing After Microfracture of Osteochondral Lesions of the Talus: A Prospective Randomized Trial. Foot Ankle Orthop. 2019 May 6;4(2):2473011419838832. doi: 10.1177/2473011419838832. eCollection 2019 Apr. PMID 35097322
- See also: VACOpaso Free OPED — http://oped.ch/vacopaso-free